CLINICAL TRIAL: NCT00872391
Title: Safety and Efficacy of Hypofractionated Stereotactic Linear Accelerator Radiotherapy of Malignant Melanoma of the Uvea
Brief Title: Hypofractionated Stereotactic Linear Accelerator Radiotherapy of Uveal Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Univ. Prof. Dr. Martin Zehetmayer, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 017/2009
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

ARMS (1):
- Hypofractionated LINAC radiotherapy (Experimental)
  Interventions: Radiation: Hypofractionated linear accelerator radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated linear accelerator radiotherapy — 10 fractions of stereotactic linear accelerator radiotherapy with 6 Gy per fraction at the 80% isodose for the planning target volume.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of hypofractionated stereotactic LINAC radiotherapy with 10 fractions at 6 Gy per fraction at the 80% isodose for the planning target volume (PTV) in patients with uveal melanoma. Patients will be followed-up for 10 years after radiotherapy regarding local tumor control, visual acuity, secondary complications and survival.

ELIGIBILITY:
Inclusion Criteria:

* The initial height of the melanoma is 7 mm or higher.
* Juxtapapillary and/or juxtamacular melanomas with a height of 3 mm or higher and if the central tumor distance to the optic disc and/or the macula is 3 mm or less.
* If other forms of conservative treatment of the melanoma are not possible.

Exclusion Criteria:

* Prior/Concomitant Treatment.
* Extrascleral tumor extension is present.
* If the presence of neovascular glaucoma is detected before treatment.
* If metastasis is detected at baseline.
* Previous participation in any study of investigational drugs within 3 month preceding day 0.
* Pregnant women are not allowed to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2009-03; Primary Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
local tumor control (tumor dimensions; secondary complications; visual acuity; survival

SECONDARY OUTCOMES:
histological assessment of the fraction of living cells in eyes requiring secondary enucleation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zehetmayer, MD, Principal Investigator — Department of Ophthalmology, Medical University of Vienna, Austria
Locations (1):
- Department of Ophthalmology and the Department of Radiotherapy and Radiobiology, Medical University of Vienna, Vienna, Vienna, Austria